CLINICAL TRIAL: NCT00620165
Title: Efficacy of Levetiracetam in Patients With Essential Tremor
Brief Title: Efficacy of Levetiracetam in Essential Tremor
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Southern California Institute for Research and Education (Other)
Responsible Party: Steven S. Schreiber, MD, Southern California Institute for Research and Education
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 00624
Record Dates: First submitted 2008-02-11; First posted 2008-02-21 (Estimated); Last update posted 2009-04-17 (Estimated); Status verified 2009-04

CONDITIONS: Essential Tremor
Keywords: tremor; writing; feeding; pouring
MeSH Terms: conditions — Essential Tremor; Tremor | interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: levetiracetam
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: levetiracetam — Subjects will receive levetiracetam titrated up over 6 weeks to a maximum dose of 3000 milligrams (mg) per day, and then continue at 1500 mg twice daily for an additional 6 weeks.
  Other Names: keppra
  Arms: 1
Drug: placebo — Subjects will receive identical placebo titrated up over 6 weeks to a maximum daily dose, and then continue twice daily for an additional 6 weeks.
  Arms: 2

SUMMARY:
Essential tremor poses one of the greatest therapeutic challenges to neurologists. This study will examine the effectiveness of the drug, levetiracetam or keppra, for the treatment of essential tremor.

DETAILED DESCRIPTION:
Currently available pharmacological treatments for essential tremor are hampered by relatively low efficacy and intolerable side effects. Recent evidence indicates that levetiracetam (LEV) may modulate the dopaminergic system. In this regard LEV has been shown to reduce L-dopa-induced dyskinesias, tardive dyskinesia and myoclonus, and is relatively well-tolerated in the elderly. Previous studies examined the efficacy of LEV for the treatment of essential tremor. However, these were either open label or relatively short duration studies. A longer term study of LEV for the treatment of essential tremor is therefore warranted. In this randomized, double-blind, placebo-controlled crossover study, ten subjects with essential tremor will be randomly assigned to receive either LEV up to a maximum dose of 3000 milligrams (mg) per day or placebo. Study drug will be titrated up over 6 weeks and continued at 1500 mg twice daily for an additional 6 weeks. Following a 4 week washout period subjects will cross over to the other arm and continued for an additional 12 weeks. Subjects will be evaluated monthly by a blinded examining neurologist and research coordinator. At each study visit subjects will receive a neurological examination and will be evaluated using a 16-item scale for tremor and medication side effects. The data derived from study drug vs. placebo groups will be compared using the Mann-Whitney U and Wilcoxon W tests.

ELIGIBILITY:
Inclusion Criteria:

* History of tremor for 5 or more years
* No other neurological problems

Exclusion Criteria:

* Prior stroke or other neurological disease, psychiatric problems
* History of renal disease
* Pregnancy

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Performance on a 16-item tremor rating scale including degree of tremor, writing, pouring and feeding. | 12 weeks per treatment arm

SECONDARY OUTCOMES:
Assessment of adverse side effects. | 12 weeks per arm

CONTACTS AND LOCATIONS:
Overall Officials: Steven S Schreiber, MD, Principal Investigator — Southern California Institute for Research and Education
Locations (1):
- VA Long Beach Healthcare System, Long Beach, California, United States